CLINICAL TRIAL: NCT03200275
Title: The Impact of Legionella Urine Antigen Testing (LUAT) on the Local Epidemiology and Diagnosis of Legionella Pneumonia - A Hospital Based Study in Malaysia
Brief Title: Impact of Legionella Urine Antigen Testing (LUAT) on the Local Epidemiology and Diagnosis of Legionella Pneumonia
Status: Completed | Type: Observational
Sponsor: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, ALBERT ANTHONY, Pulmonologist/Principal Investigator, Ministry of Health, Malaysia
Other Study IDs: NMRR-17-50-34002
Record Dates: First submitted 2017-06-24; First posted 2017-06-27 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Legionella Pneumophila Pneumonia
Keywords: Legionella urine antigen test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HOSPITALISED PNEUMONIA PATIENTS: All patients of more than 18 years of age, hospitalized consecutively for pneumonia irrespective of it being community or hospital acquired. All the patients included in this study will need to have acute symptoms of less than 2 weeks and radiological features which are compatible to pneumonia.
  They will undergo testing for Legionella pneumophila serogroup 1 urine antigen using a qualitative rapid assay following manufacturer's instructions at baseline. The diagnosis of Legionella pneumonia is made if the Immunocatch™ Legionella Urine Antigen Test is positive.
  Interventions: Diagnostic Test: Immunocatch™ Legionella Urine Antigen Test

INTERVENTIONS:
Diagnostic Test: Immunocatch™ Legionella Urine Antigen Test — A total number of 503 urine specimens from study participants will be tested with LUAT - Immunocatch™. This test utilises the immunochromatographic (ICT) membrane assay to detect antigenuria which has revolutionized the usage of UAT to diagnose Legionella infections. The results can be obtained within minutes and the test does not require any sophisticated laboratory support. A comparison of the ICT with the Enzyme Immuno Assay (EIA) test showed comparable performance characteristics.

SUMMARY:
There has never been a paper published or research done to determine the rate of Legionella species as a cause of community or nosocomial acquired pneumonia requiring hospitalization in Malaysia. Anecdotally, Legionnaires' disease is thought to be uncommon in Malaysia. This is one of the first prospective hospital-based studies to comprehensively evaluate the epidemiological and demographical factors of patients hospitalized with Legionella infection in Malaysia.

DETAILED DESCRIPTION:
Legionellosis is an environment-related, acute gram negative bacterial respiratory infection and is caused primarily by the species Legionella pneumophila, an atypical pulmonary pathogen, in the likes of mycoplasma and chlamydia species. Potentially all Legionella spp. may cause human disease, however, the majority (92%) of clinical cases are caused by L. pneumophila and the predominant serogroup is serogroup 1.

Globally, 1-5% of community acquired pneumonia patients is caused by Legionella spp. and is a challenge to public health authorities. The incidence of Legionella Pneumonia in the US has exceeded expectations and is increasing, with at least 13,000 cases occurring annually. In Singapore, Legionella spp. is responsible for 2-7% of cases of hospitalized community-acquired pneumonia.

Legionella pneumophila is being increasingly recognized as a common pathogen causing both community-acquired and nosocomial pneumonia that is responsible for significant morbidity and mortality. It is also one of the most common aetiology discovered when pneumonia is sufficiently severe to require admission to an intensive care unit. It's likely to cause a severe form of pneumonia with high likelihood of adverse medical outcomes which includes rapid deterioration, respiratory failure and the need for intensive care unit (ICU) admission.

It will be impossible to distinguish patients with Legionnaires' disease from patients with other types of pneumonia clinically. The key to diagnosis is to perform microbiologic testing when a patient is stratified into a high-risk category. Rapid diagnosis of these pneumonias is desired as delayed diagnosis and institution of appropriate antibiotics is associated with poor outcomes.

In routine clinical practice, legionellosis is rarely proven by culture whereas detection of urinary antigen is now common. In US and Europe, case detection rates were revolutionized with the usage of urine antigen test at 97% and 79% respectively. Urine antigen testing has a reported sensitivity that ranges between 76% and 86% for cases of Legionella pneumonia serogroup 1 and a specificity that approaches 100%.

In this region, urine antigen test is rarely done due to lack of clinical awareness, a perception that Legionella infection is uncommon and due to the lack of availability of this test regionally. The introduction of the immunochromatographic (ICT) membrane assay to detect antigenuria has revolutionized the usage of UAT to diagnose Legionella infections. The ICT assay is similar to a home pregnancy test and is commercially available. The test is simple to perform and does not require special laboratory equipment, and results can be obtained within 15 minutes. The investigators wish to utilize this innovation to test patients whom are hospitalized with pneumonia and determine the incidence of Legionella infection in the local setting.

ELIGIBILITY:
Inclusion Criteria:

1. More than 18 years of age,
2. Hospitalized consecutively for pneumonia irrespective of it being community or hospital acquired.
3. Acute symptoms of less than 2 weeks and radiological features which are compatible to pneumonia.

   -

Exclusion Criteria:

1. Under 18 years of age
2. Suspected/confirmed case of active tuberculosis
3. Patients who refused to give consent -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 503 patients who are consecutively hospitalised with pneumonia in Hospital Taiping from date of commencement of study.
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Legionella Pneumonia | 15 months
  The diagnosis of Legionella pneumonia is made if the Legionella Urine Antigen Test is positive. The LUAT test kit utilized in this study will not be compared to the gold standard test for Legionellosis which would be the culture on specialised media/buffered-charcoal yeast extract (BCYE) plates, as this test is not available nationwide

CONTACTS AND LOCATIONS:
Overall Officials: ALBERT IRUTHIARAJ L ANTHONY, MBBS, Principal Investigator — HOSPITAL TAIPING
Locations (1):
- Hospital Taiping, Taiping, Perak, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Touray S, Newstein MC, Lui JK, Harris M, Knox K. Legionella pneumophila cases in a community hospital: A 12-month retrospective review. SAGE Open Med. 2014 Oct 10;2:2050312114554673. doi: 10.1177/2050312114554673. eCollection 2014. PMID 26770744
- [Result] Diederen BM, Kluytmans JA, Vandenbroucke-Grauls CM, Peeters MF. Utility of real-time PCR for diagnosis of Legionnaires' disease in routine clinical practice. J Clin Microbiol. 2008 Feb;46(2):671-7. doi: 10.1128/JCM.01196-07. Epub 2007 Dec 19. PMID 18094136
- [Result] Farnham A, Alleyne L, Cimini D, Balter S. Legionnaires' disease incidence and risk factors, New York, New York, USA, 2002-2011. Emerg Infect Dis. 2014 Nov;20(11):1795-1802. doi: 10.3201/eid2011.131872. PMID 25513657
- [Result] Helbig JH, Uldum SA, Bernander S, Luck PC, Wewalka G, Abraham B, Gaia V, Harrison TG. Clinical utility of urinary antigen detection for diagnosis of community-acquired, travel-associated, and nosocomial legionnaires' disease. J Clin Microbiol. 2003 Feb;41(2):838-40. doi: 10.1128/JCM.41.2.838-840.2003. PMID 12574296
- [Result] Fiumefreddo R, Zaborsky R, Haeuptle J, Christ-Crain M, Trampuz A, Steffen I, Frei R, Muller B, Schuetz P. Clinical predictors for Legionella in patients presenting with community-acquired pneumonia to the emergency department. BMC Pulm Med. 2009 Jan 19;9:4. doi: 10.1186/1471-2466-9-4. PMID 19152698
- [Result] Levcovich A, Lazarovitch T, Moran-Gilad J, Peretz C, Yakunin E, Valinsky L, Weinberger M. Complex clinical and microbiological effects on Legionnaires' disease outcone; A retrospective cohort study. BMC Infect Dis. 2016 Feb 10;16:75. doi: 10.1186/s12879-016-1374-9. PMID 26864322
- [Result] Hollenbeck B, Dupont I, Mermel LA. How often is a work-up for Legionella pursued in patients with pneumonia? a retrospective study. BMC Infect Dis. 2011 Sep 7;11:237. doi: 10.1186/1471-2334-11-237. PMID 21899763